CLINICAL TRIAL: NCT06844903
Title: Effect of Ultrasound Acupoints on Patients With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ola Fathy Elsayed Atwa Elsharabasy, Principal Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-361
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed ultrasound at acupuncture points + Standard care program (Experimental): It will consist of 22 patients, who will receive pulsed therapeutic ultrasound (1 MHz) at bilateral acupuncture points of St29, Sp6,and unilateral acupuncture points of Ren4, Ren5, in addition to standard care program.
  Interventions: Other: Pulsed ultrasound at acupuncture points; Other: Standard care program
- Placebo ultrasound + Standard care program (Placebo Comparator): It will consist of 22 patients, who will receive placebo therapeutic ultrasound in addition to standard care program.
  Interventions: Other: Placebo ultrasound at acupuncture points; Other: Standard care program

INTERVENTIONS:
Other: Pulsed ultrasound at acupuncture points — The experimental group will receive pulsed ultrasound at bilateral acupuncture points of St29, Sp6 and unilateral acupuncture points on Ren4 and Ren5 in addition to standard care program for 12 weeks.
  Arms: Pulsed ultrasound at acupuncture points + Standard care program
Other: Placebo ultrasound at acupuncture points — The placebo group will receive the same but in Placebo manner for 12 weeks.
  Arms: Placebo ultrasound + Standard care program
Other: Standard care program — All participants in both groups will be given an info brochure, that included advice on a healthy diet as a low-carbohydrate and high-protein diet, high dietary fiber, and less saturated fat in addition to engagement in aerobic exercise, fast walking for at least 30 - 45 min, 3 days a week for 12 weeks.

SUMMARY:
This study will be conducted to evaluate the effect of ultrasound acupoints on menstrual irregularity and hormone levels on polycystic ovary syndrome (PCOS) patient.

DETAILED DESCRIPTION:
PCOS is a life-long condition and although the exact cause is yet to be identified, it is believed to have epigenetic origins. It is the main gynecological endocrinopathy of reproductive age. It is the most common cause of infertility due to anovulation. In many countries, it represents the leading cause of female infertility.

Signs and symptoms are mediated by hormonal disorder including elevated androgens and fasting insulin, and abnormal relative ratio of the gonadotropins luteinizing hormone (LH) and follicle stimulating hormone (FSH). Endocrine imbalances occur within the framework of disordered ovarian folliculogenesis, chronic anovulation, clinical signs of hyperandrogenism and metabolic syndrome.

The standard treatment of PCOS includes oral medications, lifestyle changes, and surgery. Pharmacology-based treatments are effective in only 60% of patients. Therefore, acupuncture provides an alternative.

Acupuncture therapy in female with PCOS and ovulatory disorder has been known to bring enduring useful results on the endocrine system and menstrual cycle, without complications.

In women with PCOS and IR, acupuncture was superior to metformin in improving glucose metabolism and had a lower incidence of gastrointestinal adverse effects.

There were no studies using ultrasound acupoint to improve symptoms of PCOS patients, so this study will discuss this method to describe its effect on PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults range between 18 and 35 years.
* All patients will be stopped drugs that affect the result during study period.
* body mass index (BMI) not exceeding 30 kg/m2.
* have the symptoms of oligomenorrhea or amenorrhea (appendix I).
* No documented or observable psychiatric or neurological disorders that would interfere with study participation (eg, dementia or psychosis).
* Not having any type of cancer.

Exclusion Criteria:

* Any malignancy
* Patients with severe or unstable cardiorespiratory or musculoskeletal diseases that may influence the accuracy of quantitative sensory testing results.
* Participants who refuse to stop the drugs that affect the study during study period.
* Contraindications to therapeutic ultrasound including active cancer in region of hands or feet, presence of deep vein thrombosis, complete numbness in hands or feet, metal or plastic implantation.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Serum insulin level | 12 weeks
  Blood samples will be obtained before intervention and 12 weeks after intervention by venepuncture for 20 seconds and transfer to the laboratory in gel tubes for measurement of serum insulin levels. Centrifugation will perform at 4600 rpm for 15 minutes. The Insulin Quantitative Tests are based on a solid phase enzyme-linked immunosorbent assay (ELISA). Sampling time of insulin will be an 8 -hour fasting specimen.
Serum Luteinizing Hormone (LH) level | 12 weeks
  Blood samples will be obtained before intervention and 12 weeks after intervention by venepuncture for 20 seconds and transfer to the laboratory in gel tubes for measurement of serum LH levels. Centrifugation will perform at 4600 rpm for 15 minutes. The LH Quantitative Tests are based on a solid phase enzyme-linked immunosorbent assay (ELISA). Sampling time of insulin will be an 8 -hour fasting specimen.
Serum Follicle Stimulating Hormone (FSH) level | 12 weeks
  Blood samples will be obtained before intervention and 12 weeks after intervention by venepuncture for 20 seconds and transfer to the laboratory in gel tubes for measurement of serum FSH levels. Centrifugation will perform at 4600 rpm for 15 minutes. The FSH Quantitative Tests are based on a solid phase enzyme-linked immunosorbent assay (ELISA). Sampling time of insulin will be an 8 -hour fasting specimen.
Testosterone level | 12 weeks
  Blood samples will be obtained before intervention and 12 weeks after intervention by venepuncture for 20 seconds and transfer to the laboratory in gel tubes for measurement of serum Testosterone levels. Centrifugation will perform at 4600 rpm for 15 minutes. The Testosterone Quantitative Tests are based on a solid phase enzyme-linked immunosorbent assay (ELISA). Sampling time of insulin will be an 8 -hour fasting specimen.

SECONDARY OUTCOMES:
Number of cysts on ultrasound | 12 weeks
  It will be measured before intervention and 12 weeks after intervention by ultrasonography.
Diameter of cysts on ultrasound | 12 weeks
  It will be measured before intervention and 12 weeks after intervention by ultrasonography.
Ovarian volume | 12 weeks
  It will be measured before intervention and 12 weeks after intervention by ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Fayiz Farouk El Shamy, PhD, Study Chair — Professor, Kafrelsheikh university
Locations (1):
- outpatient clinics of Mansoura Hospital, Al Mansurah, Egypt